CLINICAL TRIAL: NCT02881931
Title: FuRST 2.0: Cognitive Pre-Testing Study for a New Functional Rating Scale for Use in Huntington's Disease
Brief Title: FuRST 2.0 Cognitive Pre-Testing
Status: Completed | Type: Observational
Sponsor: CHDI Foundation, Inc. (Other)
Collaborators: Dr. Glenn T. Stebbins (Rush University Medical Center ) (Unknown); The University of Texas Health Science Center, Houston (Other); Nancy LaPelle (Unknown)
Responsible Party: Sponsor
Other Study IDs: C-000316
Record Dates: First submitted 2016-08-12; First posted 2016-08-29 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Huntington's Disease
Keywords: Huntington's disease; functional rating scale; cognitive pre-testing; patient reported outcome (PRO); HDGEC participant at Pre-Manifest stage; HDGEC participant at Early-Manifest stage; Corresponding HDGEC participant companion
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Pre-Manifest HDGEC Participant
  Interventions: Behavioral: FuRST 2.0
- Early-Manifest HDGEC Participant
  Interventions: Behavioral: FuRST 2.0
- Corresponding HDGEC participant Companion
  Interventions: Behavioral: FuRST 2.0

INTERVENTIONS:
Behavioral: FuRST 2.0 — Cognitive Pre-testing of new Functional Rating Scale

SUMMARY:
The FuRST 2.0 scale is being developed as a Patient Reported Outcome (PRO) with information coming directly from the Huntington's Disease Gene Expansion Carrier (HDGEC) and companion through self-report. The purpose of this study is to identify real or potential comprehension or usage problems with questionnaire items or response options. Through a process of structured cognitive de-briefing with HDGEC participants and companions, independently, followed by qualitative analysis, the final phrasing of the individual items and response options for the scale will be generated. Depending on the results of the first round of cognitive pre-testing, additional rounds of cognitive pre-testing may be required.

ELIGIBILITY:
Main criteria for inclusion:

1. HDGEC participant must be a participant in Enroll-HD (NCT No.: NCT01574053)
2. At least 18 years of age
3. Must be fluent in English and had his primary education in English
4. Must be willing and able to provide written informed consent

Pre-Manifest HDGECs

Criteria 1-4, and:

1. CAG length greater than or equal to 40
2. Disease Burden Score greater than or equal to 250 (calculated by the equation:

   [CAGn-35.5] X age)
3. UHDRS Diagnostic Confidence Level (DCL) < 3
4. At least five Pre-Manifest HDGEC participants should have a companion who is willing to participate in this study and complete the scale independently.

Early-Manifest (Stage 1&2) HDGECs

Criteria 1-4, and:

1. CAG length greater than or equal to 36
2. DCL=4
3. UHDRS Total Functional Capacity (TFC) ≥7
4. Participants whose companion is willing to participate in this study and complete the scale independently

Main criteria for exclusion:

1. Significant cognitive or any other impairment sufficient to interfere with study associated tasks as judged by the study Investigator or the Investigator's designee
2. Currently participating in a clinical trial involving an investigational medicinal product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants: Individuals of either gender, equal to or greater than 18 years of age. HDGEC Pre-Manifest and Early-Manifest participants (see inclusion criteria) will be recruited from English speaking Enroll-HD sites.
  Companions: Available companions for HDGEC Pre-Manifest participants will be encouraged to participate (at least five Pre-Manifest's companions are required). Companions will be identified for HDGEC Early-Manifest participants and asked to participate. Companion's participation for HDGEC Early-Manifest participant is mandatory as specified in the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2017-07-28 (Actual); Study Completion 2017-07-28 (Actual)

PRIMARY OUTCOMES:
Participants' comprehension of the FuRST 2.0 rating scale measured by qualitative analysis | 8 months
  The primary assessment will use qualitative analysis of the cognitive interview to determine the usability of the FuRST 2.0 scale in the HD population.

SECONDARY OUTCOMES:
The difference between the ratings of the HDGEC participants and the companions measured by the FuRST 2.0 rating scale | 8 months
  The secondary outcome measure will be evaluated using the Kolmogorov-Smirnov test

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - Rocky Mountain Movement Disorders Center, P.C., Englewood, Colorado
  - Hereditary Neurology Disease Centre, Inc., Wichita, Kansas
  - Columbia University, New York, New York
- CENTRE FOR MOVEMENT DISORDERS (Neuropharm Consulting), Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided